CLINICAL TRIAL: NCT00652249
Title: A Flow Monitor for Pediatric Hydrocephalic Shunts - Study of Flow Sensor With the Shunt Valve
Brief Title: Diagnosing Malfunctioning Hydrocephalic Shunt Valves With a Flow Sensor
Status: Withdrawn | Type: Observational
Why Stopped: Due to lack of enrollment.
Sponsor: Transonic Systems Inc. (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: TSI-G-HYDRO-1B-H; 2R44NS049680-02 (NIH)
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Hydrocephalus
Keywords: Hydrocephalus; shunt dysfunction; shunt flow
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Extraventricular Drainage/Pressure: Includes pediatric hydrocephalus patients that are in recovery from shunt explanation.

SUMMARY:
The study hypothesis is that a transit-time ultrasonic sensor can help doctors diagnose a malfunctioning shunt valve.

The study will simulate an implanted shunt flow monitoring system by placing the flow sensor and a programmable shunt valve into the patient's Extra-Ventricular Drainage line. Flow will be measured as the doctor raises/lowers the drainage bag to simulate the patient sitting up/lying down. The doctor will simulate a malfunctioning shunt by changing the valve's pressure release settings for each cycle of raising/lowering the bag.

By monitoring shunt flow during these changes, the doctors hope to develop new ways to diagnose malfunctioning shunt valves when implanted shunt flow monitors become available.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Hydrocephalus
* Newborn through age 20
* External Ventriculostomy with an Extra-Ventricular Drainage system installed

Exclusion Criteria:

* Not diagnosed with Hydrocephalus
* Older than age 20
* No External Ventriculostomy with an Extra-Ventricular Drainage system installed

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric hydrocephalus patients under the care of the Children's Hospital of Wisconsin, who have had an external ventriculostomy and are instrumented with an Extra-Ventricular Drainage system.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Volumetric flow of patient cerebrospinal fluid through an Extra-Ventricular Drainage System as a function of the shunt valve pressure release setting and drainage bag position. | 24 to 48 hours

SECONDARY OUTCOMES:
Recording of the pressure waveform related to the volumetric flow of patient cerebrospinal fluid through an Extra-Ventricular Drainage system. | 24 to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis J Drost, BS, MS, Principal Investigator — Transonic Systems Inc.; Bruce A Kaufman, MD, Study Director — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States